CLINICAL TRIAL: NCT01172886
Title: Metabolic Syndrome as Modifiable Risk Factor for Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sbarro Health Research Organization (Other)
Responsible Party: Sbarro Health Research Organization, Immacolata Capasso- Dept. of Senology- National Cancer Institute of Naples
Other Study IDs: icapasso
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-02

CONDITIONS: Metabolic Syndrome as Breast Cancer Risk Factor
Keywords: Metabolic Syndrome obesity visceral adiposity breast cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Healthy women and women with breast cancer have been enrolled in our nested case-control study between 2008 and 2009 in order to evaluate the association between metabolic syndrome and breast cancer, analyzing anthropometric parameters blood pressure, assessing serum HDL-C, triglyceride, fasting plasma glucose, insulin, testosterone and uric acid levels and administering a questionnaire about physical activity, food intake, tobacco use, alcohol abuse, personal and familial history of disease. Our data support the hypothesis that metabolic syndrome may be an indicator of breast cancer risk in postmenopausal women. The change of the hormonal arrangement in postmenopausal, along with an increase in visceral adiposity, probably favour the hormone dependent cell proliferation, which drives tumorigenesis. Adjustments in lifestyle with physical activity intensification and healthy diet may represent modifiable factors on which sporadic breast cancer primary prevention may work on.

DETAILED DESCRIPTION:
A total of 777 patients have been enrolled in our nested case-control study. 293 of them operated for breast cancer (cases) and 484 healthy women (controls) have been recruited between 2008 and 2009 to take part to our study for evaluating the association between MS and breast cancer. Liver or renal disease, thyroid pathology and coronary artery disease were considered exclusion criteria. After obtaining informed consent, signing the authorization to be enrolled in the study, for each woman anthropometric features were measured, including weight in kilograms, height in meters, waist and hip circumference, arterial blood pressure was taken and venous blood was collected [15]. BMI (kg/m²) was calculated from weight and height values according to World Health Organization classification (< 25 kg/m²= underweight/normal, ≥ 25 kg/m²= overweight/obese), waist and hip ratio (WHR) was obtained from waist and hip circumference, measuring the smallest circumference of both to discriminate between android and gynoid fat distribution [22]. From blood samples fasting plasma glucose, HDL-C, triglyceride, uric acid, insulin and testosterone levels were assessed. Fasting plasma glucose, HDL-C and triglyceride were measured according to NCEP ATP III criteria. The normal range for uricemia was 2.6-6.0 mg/dl. Insulin levels were defined in normal range when between 5 and 25 mcU/ml, whereas ≥ 25 mcU/ml were considered hyperinsulinemia. Testosterone levels were considered in the normal range when 0.20-1.20 ng/ml. Levels > 1.20 ng/ml were considered indicative of hyperandrogenic status. Women were asked to answer a questionnaire about chronic diseases, tobacco use, alcohol abuse, food intake, physical activity grade, parity, age of menarche, menopausal status, oral contraceptive use, hormonal therapy use, personal and familial history of cancer. According to the NCEP ATP III [10], women presenting three disorders were diagnosed with low grade MS [5], whereas women presenting more than three disorders (four or five) were diagnosed with high grade MS. Chi-squared test and logistic regression analyses (OR and 95% CI) were used to confirm the association between MS and breast cancer and to calculate the risk. Statistical significance was considered at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* healthy women
* women operated for breast cancer

Exclusion Criteria:

* Liver or renal disease,
* thyroid pathology
* coronary artery disease

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women and women operated for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 777 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Senology - National Cancer Institute of Naples, Naples, Italy, Italy